CLINICAL TRIAL: NCT03187899
Title: Superficial Cervical Plexus Blockade for Clavicle Fracture Analgesia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Principal investigator was unable to pursue research further due to time constraints.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Christopher Godlewski, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F170512002
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Pain, Postoperative; Satisfaction
Keywords: cervical plexus block; clavicle fracture; interscalene brachial plexus block
MeSH Terms: conditions — Pain, Postoperative; Personal Satisfaction | interventions — Ropivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either an interscalene brachial plexus block plus sham superficial cervical plexus block or an interscalene brachial plexus block plus a superficial cervical plexus block. The patient will be blinded as to which block they receive to prevent bias. The Attending performing/overseeing the block will not be blinded to which block is being performed. Patients receiving a traditional interscalene block and a "sham" superficial plexus block with 5-10cc of normal saline N = 20. Patients group receiving both an interscalene and a superficial plexus block N = 20.
Who Masked: Participant
Masking Description: The patient will be blinded as to which block they receive to prevent bias. The Attending performing/overseeing the block will not be blinded to which block is being performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Interscalene block plus "sham" (Sham Comparator): Patients in this group will receive a traditional interscalene block and a "sham" superficial plexus block with ropivacaine and 5-10cc of normal saline. N = 20
  Interventions: Drug: Ropivacaine; Drug: Normal saline
- Interscalene plus superficial plexus block (Active Comparator): Patients in this group will receive a traditional interscalene block and a superficial plexus block with ropivacaine . N = 20
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 0.5% of Ropivacaine will be used patients in both groups. Ropivacaine is very common in the investigator's practice of regional anesthesia. The investigator has experienced minimal adverse effects with 0.5% Ropivacaine used in volume suggested in our study.
  Other Names: Naropin
Drug: Normal saline — 5-10cc of Normal Saline will be given to patients receiving a traditional interscalene block and a sham superficial plexus block.
  Other Names: sodium chloride 0.9%
  Arms: Interscalene block plus "sham"

SUMMARY:
The goal of the study is to determine if the addition of a superficial cervical plexus block to a traditional interscalene plexus block will provide superior perioperative analgesia to an interscalene brachial plexus blockade alone for repair of clavicle fractures and non-/malunions.

DETAILED DESCRIPTION:
When patients that are possible participants in the study present for surgery, they will be offered the opportunity to participate in the trial as part of the informed consent process. Should they agree to participate, they will be randomized to receive either an interscalene + "sham" superficial cervical plexus block or an interscalene + superficial cervical plexus block. The randomization will have already been predetermined based off of envelopes that will have been created by a research assistant. Within the envelopes the proper paperwork needed to consent a participant along with a label that will be labeled either interscalene + sham superficial cervical plexus block or interscalene + superficial cervical plexus block. This will assign the randomization of each participant (this will be unknown to all study personnel until identified by the label). Their pain scores will be assessed pre-operatively as well as post-operatively .. If they are admitted to the hospital, the PI and/or Co-Investigators will assess their pain scores on a daily basis and follow-up with a phone call to assess their satisfaction with the block. Numerical pain scores (scale of 0-10) will be used to assess post-operative pain with 0 indicating no pain and 10 indicating severe pain. Post-operative pain will be assessed by compiling pain scores from 2 different sources: Numerical pain scores recorded by nursing staff (vitals section of EMR) and also pain scores ascertained by residents during rounds (progress notes). For each pain score, we will record the date and time it was obtained. If they are discharged the same day as surgery, they will receive a phone call within 48 hours to assess their pain scale and satisfaction. We will also assess nausea and vomiting, the amount and type of pain medicine they are taking, and assess if they could tell when their block wore off.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present for repair of isolated clavicle fractures and non-/malunions that consent to regional anesthesia and to be a part of the study.

Exclusion Criteria:

* Polytraumatized patients with multiple confounding injuries, patients who are not candidates for either block at the discretion of the Anesthesia Attending, patient refusal to participate in study, patient refusal of regional technique, patients with significant pulmonary disease that will not tolerate possible hemi-diaphragmatic paralysis at the discretion of the attending anesthesiologist.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain Score | baseline to 48 hours postoperatively
  Average pain score from baseline to 48 hrs postoperatively

SECONDARY OUTCOMES:
Patient Satisfaction | 48 hours postoperatively
  Patient satisfaction score at 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Godlewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No